CLINICAL TRIAL: NCT01662648
Title: An Open-label Prospective Trial to Explore the Tolerability, Safety and Efficacy of Flexibly Dosed Paliperidone ER in Subjects With Schizophrenia
Brief Title: Safety, Efficacy and Tolerability Study of Paliperidone Extended-Release (ER) in Participants With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR013534; R076477SCH3024 (Other: Janssen Pharmaceutica)
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2014-05-05 (Estimated); Status verified 2014-04

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Paliperidone; Paliperidone extended-release (ER)
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone ER: Lack of efficacy (Experimental): Paliperidone extended-release (ER) tablet in dose range of 3 to 12 milligram (mg) per day will be given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy.
  Interventions: Drug: Paliperidone ER
- Paliperidone ER: Lack of tolerability, compliance or other (Experimental): Paliperidone extended-release (ER) tablet in dose range of 3 to 12 milligram (mg) per day will be given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability, compliance or other reasons.
  Interventions: Drug: Paliperidone ER

INTERVENTIONS:
Drug: Paliperidone ER — Paliperidone extended-release (ER) tablet in dose range of 3 to 12 milligram (mg) per day will be given orally for 6 months as per Investigator's discretion.

SUMMARY:
The purpose of this study is to explore the efficacy of flexibly dosed paliperidone extended-release (ER) in participants with schizophrenia (psychiatric disorder with symptoms of emotional instability, detachment from reality, often with delusions and hallucinations, and withdrawal into the self) who were previously unsuccessfully treated with other oral antipsychotics.

DETAILED DESCRIPTION:
This is a single arm (one group of participants), multi-center, 6-month study to explore the tolerability, safety and efficacy of flexibly dosed paliperidone ER in participants with schizophrenia previously unsuccessfully treated with an oral antipsychotic medication. Antipsychotic medications are drugs that are helpful in the treatment of psychosis and have a capacity to ameliorate thought disorders. Unsuccessfully treated means that, despite the participant was treated with an adequate dose of an appropriate oral antipsychotic for an adequate period of time, previous treatment is considered unsuccessful due to lack of efficacy, lack of tolerability or safety, lack of compliance and/or other reasons. Throughout the study the investigators will adjust the dosage of each participant based on the individual needs. In general, the recommended paliperidone ER dose will be 6 milligram once daily. Participants can be either in- or outpatients and they may take their study drug with or without food. Participants who will complete this 6-month study and would like to continue will be eligible to be enrolled in an extension phase until paliperidone ER is available.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with schizophrenia
* Participant's previous treatment of schizophrenia is considered unsuccessful
* Participant is healthy on the basis of a physical examination and vital signs
* Women must be postmenopausal, surgically sterile, abstinent, or, if sexually active, agree to practice an effective method of birth control before entry and throughout the study
* Be willing and able to fill out self-administered questionnaires

Exclusion Criteria:

* Have used clozapine or Risperdal CONSTA during the last month, or have received any other conventional drug used to treat psychosis during the last 3 months
* Judged to be at high risk for adverse events, violence or self-harm
* Inability to swallow the study medication whole with the aid of water
* Pregnant or breast-feeding female
* History or current symptoms of tardive dyskinesia (involuntary movements of the facial muscles and tongue)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1117 (Actual)
Dates: Start 2007-06; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica Clinical Trial, Study Director — Janssen Pharmaceutica

RESULTS

PARTICIPANT FLOW:
Groups:
- Paliperidone ER: Lack of Efficacy: Paliperidone extended-release (ER) tablet in dose range of 3 to 12 milligram (mg) per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of efficacy.
- Paliperidone ER: Lack of Tolerability, Compliance or Other: Paliperidone extended-release (ER) tablet in dose range of 3 to 12 milligram (mg) per day was given orally for 6 months as per Investigator's discretion to participants who transitioned to Paliperidone ER from other oral antipsychotics for the main reason of lack of tolerability, compliance or other reasons.
Period: Overall Study
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Started | 520 | 597
Completed | 373 | 419
Not Completed | 147 | 178
Not completed — Death | 1 | 3
Not completed — Adverse Event | 40 | 37
Not completed — Lack of Efficacy | 17 | 16
Not completed — Participant ineligible to continue trial | 1 | 1
Not completed — Lost to Follow-up | 24 | 36
Not completed — Withdrawal by Subject | 36 | 53
Not completed — Participant non-compliant | 16 | 20
Not completed — Other | 8 | 11
Not completed — Adverse event and lack of efficacy (LOE) | 3 | 0
Not completed — LOE and other reason unspecified | 1 | 0
Not completed — LOE and Participant non-compliant | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other | Total
Number analyzed (Participants) | 520 | 597 | 1117
Age, Customized [Number; unit: Participants]
  Less than (<) 25 years | 92 (11.63) | 125 (11.90) | 217
  Greater than or equal to (>=) 25 to < 35 years | 153 | 191 | 344
  >= 35 to < 45 years | 152 | 152 | 304
  >= 45 to < 55 years | 83 | 87 | 170
  >= 55 to < 65 years | 33 | 34 | 67
  >= 65 to < 75 years | 6 | 7 | 13
  Greater than 75 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 192 | 268 | 460
  Male | 328 | 329 | 657

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 26
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: Intent to Treat (ITT) population for efficacy included all the participants who received paliperidone extended-release (ER) at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 508 | 583
units on a scale
  Baseline | 85.19 (24.97) | 65.45 (28.48)
  Week 26 | -26.60 (28.24) | -20.52 (30.05)

2. Secondary Outcome: Percentage of Participants With Greater Than or Equal to 20 Percent (%) Improvement in PANSS Total Score at Week 26
Description: The PANSS is a 30-item scale designed to assess various symptoms of schizophrenia including delusions, grandiosity, blunted affect, poor attention, and poor impulse control. The 30 symptoms are rated on a 7-point scale that ranges from 1 (absent) to 7 (extreme psychopathology). The PANSS total score consists of the sum of all 30 PANSS items and ranges from 30 to 210. Higher scores indicate worsening. Percentage of participants with greater than or equal to 20 % improvement in PANSS total score is reported here. Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Week 26
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure.
Measure: Number; unit: percentage of participants
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 508 | 583
percentage of participants | 72.83 | 71.87

3. Secondary Outcome: Change From Baseline in PANSS Total Positive Subscale Score at Week 26
Description: The Positive Subscale of PANSS (Positive and Negative Syndrome Scale) assesses seven positive-symptoms of schizophrenia. Positive symptoms refer to an excess of or distortion of normal functions. The symptoms are rated on a 7-point scale, ranging from 7 (absent) to 49 (extreme psychopathology). Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 508 | 583
units on a scale
  Baseline | 21.04 (7.15) | 15.26 (7.53)
  Week 26 | -7.17 (7.67) | -5.07 (7.88)

4. Secondary Outcome: Change From Baseline in PANSS Total Negative Subscale Score at Week 26
Description: The Negative Subscale of PANSS (Positive and Negative Syndrome Scale) assesses seven negative-symptoms of schizophrenia. Negative symptoms represent a diminution or loss of normal functions. The symptoms are rated on a 7-point scale, ranging from 7 (absent) to 49 (extreme psychopathology). Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 508 | 583
units on a scale
  Baseline | 22.73 (7.86) | 16.90 (8.13)
  Week 26 | -6.93 (7.96) | -5.32 (8.12)

5. Secondary Outcome: Change From Baseline in Clinical Global Impression-Severity (CGI-S) Score at Week 26
Description: The CGI rating scale is a 7-point global assessment that measures the clinician's impression of the severity of illness exhibited by a participant. A rating of 1 indicates to "normal, not at all ill" and a rating of 7 indicates "among the most extremely ill participants". Higher scores indicate worsening. Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 508 | 583
units on a scale
  Baseline | 4.24 (0.83) | 3.29 (1.12)
  Week 26 | -1.12 (1.28) | -0.98 (1.30)

6. Secondary Outcome: Change From Baseline in Personal and Social Performance (PSP) Scale at Week 26
Description: The PSP scale assesses the degree of dysfunction within 4 domains of behavior: socially useful activities, personal and social relationships, self-care and disturbing and aggressive behavior. The score ranges from 1 to 100, divided into 10 equal intervals to rate the degree of difficulty (1, absent to 6, very severe) in each of the 4 domains. Participants with a score of 71 to 100 have a mild degree of difficulty; from 31 to 70, varying degrees of disability; less or equal to 30, functioning so poorly as to require intensive supervision. Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment. "N" (number of participants analyzed) signifies the participants evaluable for this measure and 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 506 | 583
units on a scale
  Baseline (n= 506, 583) | 55.07 (15.68) | 66.03 (15.65)
  Week 26 (n= 501, 574) | 13.76 (17.80) | 11.14 (17.53)

7. Secondary Outcome: Change From Baseline in Sleep Quality at Week 26
Description: Sleep quality was assessed by an 11-point visual analog scale that rates how well participants sleep. Participants indicated on the scale (from 0 to 100 millimeter) how well they have slept in the previous 7 days (from 0: "very badly" to 100: "very well"). Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 507 | 581
millimeter (mm)
  Baseline (n= 507, 581) | 63.53 (27.37) | 67.40 (27.13)
  Week 26 (n= 504, 574) | 11.57 (35.70) | 8.19 (35.93)

8. Secondary Outcome: Change From Baseline in Daytime Drowsiness at Week 26
Description: Daytime Drowsiness was assessed by an 11-point visual analog scale that rates how well participants sleep. Participants indicated on the scale (from 0 to 100 millimeter) how often they have felt drowsy within the previous 7 days (from 0: "not at all" to 100:"all the time"). Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: millimeter (mm)
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 507 | 581
millimeter (mm)
  Baseline (n= 507, 581 ) | 32.80 (27.56) | 34.54 (28.61)
  Week 26 (n= 504, 574) | -9.52 (32.29) | -11.54 (34.53)

9. Secondary Outcome: Number of Participants Within Each Category of Patient Satisfaction Score
Description: Participants were interviewed at baseline and at the end of the trial (Week 26) to assess their satisfaction with the current treatment on a 5-point scale (very good, good, reasonable, moderate or poor). Data for two groups is presented here, based on the reason to switch: lack of efficacy and lack of tolerability, compliance or other who switched from other previous antipsychotic drugs to paliperidone.
Time Frame: Baseline and Week 26
Population: ITT population for efficacy included all the participants who received paliperidone ER at least once and who had at least 1 post baseline efficacy assessment."N" (number of participants analyzed) signifies participants evaluable for this measure and "n" signifies those participants who were evaluated for this measure at specified time point.
Measure: Number; unit: participants
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Number analyzed (Participants) | 507 | 583
participants
  Very Good: Baseline (n= 507, 583) | 8 (32.74) | 21 (34.67)
  Good: Baseline (n= 507, 583) | 74 | 151
  Reasonable: Baseline (n= 507, 583) | 256 | 305
  Moderate: Baseline (n= 507, 583) | 158 | 97
  Poor: Baseline (n= 507, 583) | 11 | 9
  Very Good: Week 26 (n=492, 563) | 120 | 156
  Good: Week 26 (n=492, 563) | 173 | 253
  Reasonable: Week 26 (n=492, 563) | 112 | 94
  Moderate: Week 26 (n=492, 563) | 70 | 50
  Poor: Week 26 (n=492, 563) | 17 | 10

ADVERSE EVENTS:
Time Frame: 26 weeks
Description: Safety population included all the participants who received paliperidone extended-release (ER) at least once and provided any post-baseline information.
Arm/Group | Paliperidone ER: Lack of Efficacy | Paliperidone ER: Lack of Tolerability, Compliance or Other
Serious Adverse Events (participants affected / at risk) | 35/512 | 29/587
Other Adverse Events (participants affected / at risk) | 208/512 | 239/587
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER: Lack of Efficacy (N=512) | Paliperidone ER: Lack of Tolerability, Compliance or Other (N=587)
Schizophrenia (Psychiatric disorders) | 12 | 7
Psychotic disorder (Psychiatric disorders) | 7 | 3
Aggression (Psychiatric disorders) | 1 | 2
Agitation (Psychiatric disorders) | 2 | 1
Hallucination (Psychiatric disorders) | 1 | 1
Suicidal behaviour (Psychiatric disorders) | 1 | 1
Abnormal behaviour (Psychiatric disorders) | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0
Delusion of grandeur (Psychiatric disorders) | 0 | 1
Grandiosity (Psychiatric disorders) | 1 | 0
Hallucination, auditory (Psychiatric disorders) | 0 | 1
Hostility (Psychiatric disorders) | 1 | 0
Mania (Psychiatric disorders) | 0 | 1
Schizoaffective disorder (Psychiatric disorders) | 0 | 1
Schizophrenia, disorganized type (Psychiatric disorders) | 0 | 1
Extrapyramidal disorder (Nervous system disorders) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Akathisia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Dystonia (Nervous system disorders) | 1 | 0
Poor quality sleep (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Investigation (Investigations) | 1 | 2
Weight decreased (Investigations) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
(General disorders) | 0 | 2
Cardiac arrest (Cardiac disorders) | 0 | 1
Oculogyration (Eye disorders) | 1 | 0
Poisoning (Injury, poisoning and procedural complications) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Drowning (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Convulsion (Nervous system disorders) | 1 | 0
Acute psychosis (Psychiatric disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Blood pressure increased (Investigations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone ER: Lack of Efficacy (N=512) | Paliperidone ER: Lack of Tolerability, Compliance or Other (N=587)
Extrapyramidal disorder (Nervous system disorders) | 34 | 21
Headache (Nervous system disorders) | 23 | 24
Dizziness (Nervous system disorders) | 16 | 22
Akathisia (Nervous system disorders) | 13 | 18
Somnolence (Nervous system disorders) | 9 | 20
Tremor (Nervous system disorders) | 9 | 12
Parkinsonism (Nervous system disorders) | 0 | 6
Poor quality sleep (Nervous system disorders) | 9 | 0
Insomnia (Psychiatric disorders) | 50 | 68
Restlessness (Psychiatric disorders) | 9 | 13
Anxiety (Psychiatric disorders) | 0 | 9
Psychotic disorder (Psychiatric disorders) | 9 | 0
Depression (Psychiatric disorders) | 0 | 6
Nausea (Gastrointestinal disorders) | 17 | 23
Vomiting (Gastrointestinal disorders) | 15 | 16
Salivary hypersecretion (Gastrointestinal disorders) | 0 | 7
Constipation (Gastrointestinal disorders) | 8 | 8
Pyrexia (General disorders) | 0 | 9
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 8
Weight increased (Investigations) | 0 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 6
Amenorrhoea (Reproductive system and breast disorders) | 0 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 6
Oculogyration (Eye disorders) | 0 | 6
Palpitations (Cardiac disorders) | 6 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No